CLINICAL TRIAL: NCT05350098
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Plant-protein Diets in Patients With Chronic Kidney Disease: a Pilot-study
Brief Title: Efficacy of Plant-protein Diets in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Osaka University (Other)
Responsible Party: Principal Investigator, Yusuke Sakaguchi, assistant professor, Osaka University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21371
Record Dates: First submitted 2022-04-06; First posted 2022-04-27 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Disease Stage 5
Keywords: plant-protein diets; chronic kidney disease; uremic solutes; metabolic acidosis; chronic kidney disease-mineral and bone disorder; gut microbiome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A dietary intervention of plant-protein based diets (Experimental)
  Interventions: Other: Plant-protein Diets
- A dietary intervention of control diets (Active Comparator)
  Interventions: Other: Control Diets

INTERVENTIONS:
Other: Plant-protein Diets — Participants will consume meals with 70% plant-based protein three times a day. Participants will be prohibited to have meals other than experimental diets and to drink milk and soy milk.
  Arms: A dietary intervention of plant-protein based diets
Other: Control Diets — Participants will consume meals with 50% plant-based protein three times a day. Participants will be prohibited to have meals other than experimental diets and to drink milk and soy milk.
  Arms: A dietary intervention of control diets

SUMMARY:
The purpose of this study is to evaluate the efficacy of plant-protein diets for 12 weeks in patients with advanced chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. patients with chronic kidney disease who were referred to the Outpatient Department of Nephrology at Osaka University Hospital
2. eGFR < 20 mL/min/1.73 m2
3. taking anigiotensin-converting enzyme inhibitors or angiotensin Ⅱ receptor blockers or angiotensin receptor neprilysin inhibitor
4. K < 5.5 mEq/L

Exclusion Criteria:

1. Being planned to intitate renal replacement therapies within 3 months
2. Having inflammatory bowel diseases
3. History of gastrointestinal tract surgery
4. Taking antibiotics within 1 month before the entry
5. Taking or being planned to start warfarin
6. Having dietary allergies
7. Having difficulty in oral intake
8. During pregnancy or breastfeeding
9. Unsuitable for participant in the trial by an attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in serum levels of indoxyl sulfate, p-Cresyl sulfate and trimethylamine N-Oxide | 4 weeks after starting intervention

SECONDARY OUTCOMES:
Change in eGFR | 4 weeks after starting intervention
Change in urinary protein creatinine ratio | 4 weeks after starting intervention
Change in serum bicarbonete levels | 4 weeks after starting intervention
Change in urinary citrate to creatinine ratio | 4 weeks after starting intervention
  The measurement of this outcome was abandoned because of the end of sales for its measuring reagent (F-kit citrate; JK International, Tokyo, Japan) in Japan on December 23, 2022. This decision had been made before we initiatited the recruitement of study participants.
Change in blood pressure | 4 weeks after starting intervention
Change in serum levels of calcium, phosphate, intact parathyroid hormone and intact fibroblast growth factor 23 | 4 weeks after starting intervention
Change in serum levels of acetic acid, propionic acid and butyric acid | 4 weeks after starting intervention
Diversity and composition of the gut microbiota | 4 weeks after starting intervention
Change in muscle mass | 4 weeks after starting intervention
Dietary adherence | 4 weeks after starting intervention
  How many times participants have the study diet during the study period.
The number of oral medications including antihypertensive drugs, diuretics, potassium tablets, potassium binders, phosphate binders, calcium tablets, active vitamin D3 analogs and sodium bicarbonate | 4 weeks after starting intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Osaka University, Suita, Osaka, Japan